CLINICAL TRIAL: NCT04804995
Title: Headache in Ramadan.
Brief Title: Investigating the Frequency and Phenotype of Headaches Associated With Fasting During the Month of Ramadan.
Status: Completed | Type: Observational
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Mohammad Al-Mahdi Al-Karagholi, MD, Danish Headache Center
Other Study IDs: Ramadan2021
Record Dates: First submitted 2021-03-16; First posted 2021-03-18 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Headache; Migraine
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heathy participants
  Interventions: Other: There is no intervention.
- migraine patients
  Interventions: Other: There is no intervention.

INTERVENTIONS:
Other: There is no intervention. — No intervention.

SUMMARY:
Headaches are more common in the month of Ramadan in patients who already suffer from migraine. The object of the present study is investigate the frequency in the Ramadan month .

ELIGIBILITY:
Inclusion Criteria:

* age 18-60 years.
* expectation of fasting for at least 21 of 30 days during the month of Ramadan.
* understand and answer the questionnaire sent out in Danish.

Exclusion Criteria:

* non-compliance with the headache calendar (defined as non-registration of at least 21 days per 30 days).

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: Healthy participants and migraine patients.
Sampling Method: Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Headache frequency | Daily headache diary in three months.
  The frequency of headaches is higher in the first half of Ramadan month compared to the last half.
Headache frequency | Daily headache diary in three months.
  The frequency of headaches is higher in the month before Ramadan compared to the month after ramadan.

CONTACTS AND LOCATIONS:
Overall Officials: Faisal Mohammad Amin, Principal Investigator — Danish Headache Center
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No